CLINICAL TRIAL: NCT04337671
Title: Impact of Aerobic Training on Sleep Quality and Aerobic Fitness in Male Patients With Pulmonary Artery Hypertension: a Randomized Control Study
Brief Title: Impact of Aerobic Training on Sleep Quality and Aerobic Fitness in Male Patients With Pulmonary Artery Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba Ahmed Ali Abdeen, Assistant Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2019HAHA
Record Dates: First submitted 2020-03-31; First posted 2020-04-08 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Pulmonary Artery Hypertension
MeSH Terms: conditions — Familial Primary Pulmonary Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training group (A) (Experimental): The training was a moderate intensity aerobic training on a bicycle ergo-meter(corresponding to 60% to 70% of the maximal heart rate they reach during peak oxygen uptake in the initial exercise test) for 30 to 45 min/day, 3 sessions/week for 12 weeks (36 sessions). In addition to their prescribed medications.
  Interventions: Other: Moderate intensity aerobic training
- control group (B) (No Intervention): Control group not receiving any training . They are taking their prescribed medications only.

INTERVENTIONS:
Other: Moderate intensity aerobic training — The exercise program consisted of 5 minutes warm-up, 15-30 minutes of moderate aerobic exercises and 10 minutes cool-down, respectively.
  Frequency: 3 sessions/week , and Duration:12 weeks.
  Arms: Training group (A)

SUMMARY:
This study investigated the effect of 12 weeks of aerobic training on sleep quality and aerobic fitness in patients with Pulmonary arterial hypertension(PAH).

DETAILED DESCRIPTION:
Thirty male PAH patients were included in the study. They were randomized into two equal groups; Training group (A) and Control group(B). Right ventricular systolic pressure (RVSP) measured using Doppler Echocardiography , Pittsburg sleep quality index (PSQI) questionnaire with the wrist worn actigraph used for the assessment of sleep disturbance, and Cardiopulmonary exercise testing (CPET) measurements included maximal heart rate and VO2max .All were measured before and after the study period for both groups.The training was a moderate intensity aerobic training on a bicycle ergometer (corresponding to 60% to 70% of the maximal heart rate they reach during peak oxygen uptake in the initial exercise test) for 30 to 45 min/day, 3 sessions/week for 12 weeks (36 sessions).

ELIGIBILITY:
Inclusion Criteria:

* Patients who were clinically stable and compensated under optimized medical therapy
* World health organization (WHO) Classification of functional class II to III PAH
* Patients with ejection fraction ≥ 40%
* Non-smokers
* body mass index ≤ 35 kg/m2

Exclusion Criteria:

* Any patient with respiratory failure
* unstable angina
* renal, hepatic or neuromuscular disorders
* history of syncopal attacks
* uncontrolled systemic hypertension
* peripheral vascular disease
* serious cardiac dysrhythmias on resting ECG
* evidence of severe COPD at pulmonary function testing,
* any known musculoskeletal or neurological conditions that might interfere with the execution or the assessment of the exercise

Ages: 45 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males are selected because the functional capacity parameters measured maximum oxygen consumption(VO2 max) differs from males and females as it relies on body compostion , body size, amount of muscle mass and also on ventilatory parameters
Enrollment: 30 (Actual)
Dates: Start 2018-06-02 (Actual); Primary Completion 2019-11-29 (Actual); Study Completion 2019-12-28 (Actual)

PRIMARY OUTCOMES:
Pulmonary artery systolic pressure (PASP) | change from baseline at 12 weeks
  Pulsed Doppler Echocardiogram for assessing PASP as calculated from the gradient across the tricuspid valve using the modified Bernoulli equation.
Subjective self-report questionnaire that assesses sleep quality | change from baseline at 12 weeks
  The Pittsburgh Sleep Quality Index is a subjective self-report questionnaire that assesses sleep quality over a 1-month time interval in different populations It is 5 points score (0 means normal, 5 means severe sleep disturbance)
Determining sleep patterns | change from baseline at 12 weeks
  Determining sleep patterns by using actigraph to assess suspected certain sleep disorders,
Measuring aerobic fitness | change from baseline at 12 weeks
  Level of aerobic fitness assessed by using Cardiopulmonary exercise testing (CPET) through incremental exercise intensity until voluntary exhaustion.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Atef H, Abdeen H. Effect of exercise on sleep and cardiopulmonary parameters in patients with pulmonary artery hypertension. Sleep Breath. 2021 Dec;25(4):1953-1960. doi: 10.1007/s11325-020-02286-9. Epub 2021 Feb 18. PMID 33604801